CLINICAL TRIAL: NCT00002624
Title: VIDEO ASSISTED WEDGE RESECTION (VAR) AND RADIOTHERAPY FOR HIGH RISK T1 NON-SMALL CELL LUNG CANCER: A PHASE II STUDY
Brief Title: Video-Assisted Surgery Followed by Radiation Therapy in Treating Patients With Stage I Non-small Cell Lung Cancer and Poor Heart and Lung Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9335; U10CA031946 (NIH); CDR0000063987 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Chemotherapy, Adjuvant; Video-Assisted Surgery; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiotherapy + surgery (Experimental): Patients begin radiotherapy 2-8 weeks postoperatively. Patients with complete resection undergo radiotherapy 5 days a week for 5.6 weeks. Patients with incomplete resection undergo radiotherapy 5 days a week for 6.6 weeks.
  Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.
  Interventions: Procedure: adjuvant therapy; Procedure: diagnostic thoracoscopy; Procedure: therapeutic thoracoscopy; Procedure: video-assisted surgery; Radiation: radiation therapy

INTERVENTIONS:
Procedure: adjuvant therapy
Procedure: diagnostic thoracoscopy
Procedure: therapeutic thoracoscopy
Procedure: video-assisted surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Video-assisted surgery followed by radiation therapy may be an effective treatment in patients whose poor heart and lung function make them high risk for standard surgery.

PURPOSE: Phase II trial to study the effectiveness of video-assisted surgery followed by radiation therapy in treating patients with stage I non-small cell lung cancer and poor heart and lung function.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of video-assisted thoracoscopic wedge resection (VAR) followed by radiotherapy in patients with stage I non-small cell lung cancer and cardiopulmonary dysfunction.
* Determine the incidence of locoregional recurrence in patients treated with this regimen.
* Determine the overall and disease-free survival in patients treated with this regimen.
* Determine the technical feasibility of ipsilateral lymph node sampling and complete resection with VAR in these patients.
* Determine the incidence of conversion to open thoracotomy in these patients.
* Determine the short- and long-term complications associated with VAR in these patients.
* Determine the toxicity of adjuvant radiotherapy after VAR in these patients.

OUTLINE: This is a multicenter study.

Patients undergo video-assisted thoracoscopic wedge resection. Surgeons attempt sampling and identification of all ipsilateral, mediastinal, and hilar lymph nodes. When accessible, lobar lymph nodes must also be sampled. If the tumor margins are positive, further resection of the margins must be attempted. Open thoracotomy may be required for technical reasons.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Known or suspected, single, peripheral, stage T1 N0 M0 lung tumor

  * Tumor must not be identifiable by bronchoscopy

    * Bronchoscopically visible cancer or bronchial distortions considered related to tumor
  * Positive cytology by bronchoscopy allowed if no gross abnormality visible
  * Mediastinoscopy required for nodes greater than 1 cm
  * No pleural effusions
  * No metastatic or N2 disease on CT scan
  * Lesion must be accessible for video-assisted thoracoscopic wedge resection
* High cardiopulmonary risk for thoracotomy with at least 1 of the following criteria:

  * FEV1 less than 40% predicted
  * DLCO less than 50% predicted
  * Supplemental oxygen requirement
  * Chronic PaCO2 greater than 45 mm Hg
  * Maximum oxygen consumption (VO2 max) less than 15 mL/kg/min
* Patients who appear at high risk for non-pulmonary reasons (e.g., patients who are elderly or with renal or cardiac failure) may be eligible only if VO2 max or other criteria above are met
* Eligible for radiotherapy after completion of wedge resection if histologic documentation of non-small cell lung cancer, including any of the following subtypes:

  * Squamous cell carcinoma
  * Adenocarcinoma
  * Bronchoalveolar cell
  * Large cell anaplastic carcinoma
* Cytology from bronchial washings and transthoracic needle aspiration not acceptable

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* 0-2

Other:

* No other malignancy within the past 5 years except nonmelanomatous skin cancer or carcinoma in situ of the cervix
* Weight loss no greater than 10% within the past 6 months

PRIOR CONCURRENT THERAPY:

Radiotherapy

* No prior thoracic irradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 1994-12; Primary Completion 2005-04 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility of video-assisted thoracoscopic wedge resection (VAR) | Up to 10 years
Determine the incidence of locoregional recurrence in patients treated with this regimen | Up to 10 years
Determine the overall and disease-free survival | Up to 10 years
Determine the short- and long-term complications associated with VAR in these patients | Up to 10 years
Determine the technical feasibility of ipsilateral lymph node sampling and complete resection with VAR in these patients | Up to 10 years
Determine the toxicity of adjuvant radiotherapy after VAR in these patients | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Hani Shennib, MD, Study Chair — Montreal General Hospital
Locations (16):
- United States (13):
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center-Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Midlands Cancer Center at Midlands Community Hospital, Papillion, Nebraska
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University Hospital, Philadelphia, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
- Westmead Hospital, Westmead, New South Wales, Australia
- Instituto de Enfermedades Neoplasicas, Lima, Peru
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Result] Shennib H, Bogart J, Herndon JE, Kohman L, Keenan R, Green M, Sugarbaker D; Cancer and Leukemia Group B; Eastern Cooperative Oncology Group. Video-assisted wedge resection and local radiotherapy for peripheral lung cancer in high-risk patients: the Cancer and Leukemia Group B (CALGB) 9335, a phase II, multi-institutional cooperative group study. J Thorac Cardiovasc Surg. 2005 Apr;129(4):813-8. doi: 10.1016/j.jtcvs.2004.05.011. PMID 15821648
- [Result] Bogart J, Shennib H, Kohman L, et al.: Radiotherapy following thorascopic wedge resection (TWR) of T1 non-small cell lung cancer (NSCLC) in high risk patients: a Cancer and Leukemia Group B and Eastern Cooperative Oncology Group Phase II Trial. [Abstract] Proceedings of the American Society of Clinical Oncology 19: A1907, 2000.